CLINICAL TRIAL: NCT06693869
Title: The Risk of Surgical Cancellation in Adult Patients Assessed by Telephone Versus In-person for Scheduled Non-cardiac Elective Surgery.
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2024
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Surgical Procedures; Telemedicine; Preanesthetic Medication; Preoperative Care; Anesthesia; Risk Assessment; Postoperative Complications; Noncardiac Surgery; Elective Surgery Cancellation
Keywords: Surgical Cancellation Risk; Preanesthetic Assessment; Telephone Preoperative Evaluation; In-Person Preoperative Evaluation; Elective Non-Cardiac Surgery; Surgery Cancellation Rate; Preanesthetic Evaluation Telemedicine; Telehealth in Preoperative Care; Comparison of Preanesthetic Methods; Risk Assessment for Surgery Cancellation; Postoperative Complications in Non-Cardiac Surgery; Patient Satisfaction with Telemedicine; Perioperative Outcomes; Remote Preoperative Consultation; Surgical Risk Management; Telemedicine vs. In-Person Evaluation; Retrospective Study in Anesthesiology; Surgical Outcome Prediction; Telemedicine in Anesthesiology; Preanesthetic Teleconsultation
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Telephone pre-anesthetic evaluation: Surgical patients scheduled for elective non-cardiac surgery underwent pre-anesthetic evaluation through a telephone consultation, which included a review of medical history, medications, and risk factors made by anesthesiologists. No physical examination was conducted.
- In-Person pre-anesthetic evaluation: Surgical patients scheduled for elective non-cardiac surgery received an in-person pre-anesthetic evaluation performed by an anesthesiologist, which included a physical examination and a thorough risk assessment.

SUMMARY:
Telemedicine has been regulated in Colombia since 2006, with applications in anesthesia being explored since 2004 to improve accessibility and reduce costs. Although Decree 538 of 2020 expanded telemedicine's medical applications, challenges such as connectivity issues and the need for training remain. Telemedicine has shown promise in rural areas of Colombia, particularly for managing chronic diseases. However, further evidence is needed regarding the effectiveness of telephone pre-anesthetic evaluations.

This study aims to investigate the implementation of telephone assessments for non-cardiac surgery and their impact on surgical cancellations compared to in-person pre-anesthetic evaluations. The primary question we seek to answer is:

Does telephone pre-anesthetic assessment in non-cardiac surgical patients carry a higher risk of surgical cancellations compared to in-person evaluations?

To address this question, we will evaluate patients' medical records in two hospitals where patients were assessed using both telephone and in-person modalities.

DETAILED DESCRIPTION:
The COVID-19 pandemic accelerated the adoption of telemedicine, including its application in preoperative anesthesia evaluations. While the use of telephone assessments in anesthesiology is increasing, there is ongoing debate about their accuracy in identifying medical risks and predicting potential post-surgical outcomes. Preanesthetic evaluations are essential for determining patient suitability for surgery and for classifying surgical risk.

Despite the benefits of increased accessibility and cost reduction associated with telephone assessments, concerns persist regarding their ability to match the thoroughness of in-person evaluations. This is particularly relevant given the potential for higher surgical cancellation rates.

In Colombia, telephone preanesthetic evaluations for non-cardiac elective surgeries are a recent development, potentially optimising resource use and enhancing patient satisfaction. However, it is crucial to investigate whether they result in a cancellation rate comparable to in-person assessments, as this could be a significant barrier to widespread implementation. This study examines the effectiveness of telephone assessments for non-cardiac surgeries and their impact on surgical cancellations compared to in-person preanesthetic evaluations. A secondary objective of the study is to evaluate the incidence of perioperative complications, including cardiovascular issues, pulmonary complications, bleeding, unexpected ICU admissions, and non-anticipated difficult airways.

ELIGIBILITY:
Inclusion Criteria:

- Patients who were scheduled for elective non-cardiac surgery.

Exclusion Criteria:

* Pregnant patients.
* More than three months between the pre-anesthetic evaluation and the scheduled surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults aged 18 years and older scheduled for ambulatory elective non-cardiac surgeries at two healthcare institutions: Alma Mater Hospital of Antioquia and San Vicente Fundación University Hospital in Medellín.
Sampling Method: Non-Probability Sample
Enrollment: 1180 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Surgical cancellation incidence | Pre-surgery
  The incidence of surgical procedure cancellation because of a medical condition affecting the patient and the surgery.

SECONDARY OUTCOMES:
Incidence of unanticipated difficult airway | During the surgery
  Incidence of difficulties with facemask ventilation of the upper airway, tracheal intubation, or both.
Incidence of perioperative cardiovascular complications | Late postoperative (until 7 days after surgery)
  Incidence of any perioperative cardiovascular complications during intraoperative or postoperative periods: all-cause death, sudden cardiac arrest, congestive heart failure, non-fatal myocardial infarction (MI), pulmonary embolism.
Incidence of postoperative mechanical ventilation | early postoperative (until 2 hours after surgery)
  Incidence of postoperative mechanical ventilation.
Incidence of perioperative respiratory complications | Late postoperative (until 7 days after surgery)
  The occurrence of respiratory complications in the perioperative period, including pneumonia, can happen within seven days following surgery
Incidence of unplanned ICU admission | early postoperative (until 2 hours after surgery)
  Incidence of unplanned ICU admission in the postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Fabian D Casas, Professor, Study Director — Universidad de Antioquia
Locations (1):
- University of Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muñoz L, Reyes LE, Infante S, Quiroga J, Cabrera L, Obando N, et al. Cancelación de procedimientos electivos y su relación con la valoración preanestésica. Rev Repert Med Cir. 17 de abril de 2018;27(1):24-9.
- [Background] Thompson T, Brophy T, Modgil V, Pearce I. Remote healthcare consultations: the new era of outpatient medicine. Trends Urol Mens Health. 2020;11(5):25-8.
- [Background] Ryu S. Telemedicine: Opportunities and Developments in Member States: Report on the Second Global Survey on eHealth 2009 (Global Observatory for eHealth Series, Volume 2). Healthc Inform Res. junio de 2012;18(2):153-5.
- [Background] Prados Castillejo JA. [Telemedicine, also a tool for the family doctor]. Aten Primaria. 2013 Mar;45(3):129-32. doi: 10.1016/j.aprim.2012.07.006. Epub 2012 Sep 11. No abstract available. Spanish. PMID 22981128
- [Background] Castillo VS, Cano CAG, Gonzalez-Argote J. Telemedicine and mHealth Applications for Health Monitoring in Rural Communities in Colombia: A Systematic Review.
- [Background] Aldawoodi NN, Muncey AR, Serdiuk AA, Miller MD, Hanna MM, Laborde JM, Garcia Getting RE. A Retrospective Analysis of Patients Undergoing Telemedicine Evaluation in the PreAnesthesia Testing Clinic at H. Lee Moffitt Cancer Center. Cancer Control. 2021 Jan-Dec;28:10732748211044347. doi: 10.1177/10732748211044347. PMID 34644199
- [Background] Wongtangman K, Azimaraghi O, Freda J, Ganz-Lord F, Shamamian P, Bastien A, Mirhaji P, Himes CP, Rupp S, Green-Lorenzen S, Smith RV, Medrano EM, Anand P, Rego S, Velji S, Eikermann M. Incidence and predictors of case cancellation within 24 h in patients scheduled for elective surgical procedures. J Clin Anesth. 2022 Dec;83:110987. doi: 10.1016/j.jclinane.2022.110987. Epub 2022 Oct 26. PMID 36308990
- [Background] Zhang K, Rashid-Kolvear M, Waseem R, Englesakis M, Chung F. Virtual preoperative assessment in surgical patients: A systematic review and meta-analysis. J Clin Anesth. 2021 Dec;75:110540. doi: 10.1016/j.jclinane.2021.110540. Epub 2021 Oct 11. PMID 34649158
- [Background] Schmidt AP, Modolo NSP, de Amorim CG, Simoes CM, Kraychete DC, Joaquim EHG, Lineburger EB, Papa FV, Fernandes FC, Mendes FF, Guimaraes GMN, Barros GAM, Silva-Jr JM, Navarro E Lima LH, Azi LMTA, Carvalho LIM, Stefani LC, Garcia LV, Malbouisson LMS, Salgado-Filho MF, Nascimento Junior PD, Alves RL, Carvalho VH, Quintao VC, Carmona MJC. Two years of the COVID-19 pandemic: an anesthesiology perspective. Braz J Anesthesiol. 2022 Mar-Apr;72(2):165-168. doi: 10.1016/j.bjane.2022.02.004. Epub 2022 Feb 19. No abstract available. PMID 35189166
- [Background] Kamdar NV, Huverserian A, Jalilian L, Thi W, Duval V, Beck L, Brooker L, Grogan T, Lin A, Cannesson M. Development, Implementation, and Evaluation of a Telemedicine Preoperative Evaluation Initiative at a Major Academic Medical Center. Anesth Analg. 2020 Dec;131(6):1647-1656. doi: 10.1213/ANE.0000000000005208. PMID 32841990
- [Background] Lozada MJ, Nguyen JT, Abouleish A, Prough D, Przkora R. Patient preference for the pre-anesthesia evaluation: Telephone versus in-office assessment. J Clin Anesth. 2016 Jun;31:145-8. doi: 10.1016/j.jclinane.2015.12.040. Epub 2016 Apr 15. PMID 27185698
- [Background] Garg R, Hoda W. Emergence of Telehealth for anesthesiologists in COVID-19-boon for all! J Anaesthesiol Clin Pharmacol. 2020 Jul-Sep;36(3):417-419. doi: 10.4103/joacp.JOACP_416_20. Epub 2020 Sep 29. No abstract available. PMID 33487917